CLINICAL TRIAL: NCT04926363
Title: Prevalence of Cardiovascular Risk Factors in People With Upper Vestibular Neuritis
Brief Title: Prevalence of Cardiovascular Risk Factors in Upper Vestibular Neuritis
Acronym: NEVRITE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7665
Record Dates: First submitted 2021-06-04; First posted 2021-06-15 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-06

CONDITIONS: Vestibular Neuritis
Keywords: Vestibular neuritis; Anterior vestibular artery
MeSH Terms: conditions — Vestibular Neuronitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vestibular neuritis is the second cause of vertigo, it constitutes 5 to 6% of the aetiologies of vertigo in an otoneurological consultation.

Infection or reactivation of a neurotropic virus of the herpes group (HSV-1) in the vestibular lymph node is thought to be the cause of the unilateral vestibular deficit.

Upper vestibular neuritis is more common than lower, or total involvement. Goebel (2) explains this by an anatomical predisposition of the vestibular nerve canal to inflammation, unlike the singular nerve canal which is shorter and wider giving way to a certain degree of edema without consequence on its contents.

However, the innervation territory of the superior vestibular nerve is superimposable on the territory supplied by the anterior vestibular artery. The anterior, lateral semicircular canals and the utricle are affected. Current complementary vestibular and imaging examinations cannot differentiate between inflammatory or vascular involvement in upper vestibular neuritis.

The increased presence of cardiovascular risk factors in patients with upper vestibular neuritis would be an argument in favor of ischemic involvement of the anterior vestibular artery.

ELIGIBILITY:
nclusion criteria:

* Major subject (≥18 years old),
* Subject having presented an episode of upper vestibular neuritis recorded on the Video Head Impulse Test Ulmer device at the HUS between 01/01/2016 and 01/31/2020,
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Patient who expressed his opposition to participating in the study,
* Total vestibular neuritis,
* impossibility of providing the subject with enlightened information (difficulties in understanding the subject, etc.)
* Subject under safeguard of justice,
* Subject under guardianship or guardianship,
* Lack of video head impulse test data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major having presented an episode of upper vestibular neuritis recorded on the Video Head Impulse Test Ulmer device at the HUS between 01/01/2016 and 01/31/2020,
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-04 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of cardiovascular risk factors in people with upper vestibular neuritis | Files analysed retrospectively from January 01, 2016 to January 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Anne CHARPIOT, MD, PhD, Study Director — Service ORL et de CCF- Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service ORL et de CCF - Hôpitaux Universitaires de Strasbourg, Strasbourg, France